CLINICAL TRIAL: NCT05560139
Title: The Effect of Transcranial Direct Current Stimulation on Fatigue Among Multiple Sclerosis Patients
Brief Title: The Effect of Transcranial Direct Current Stimulation on Fatigue Among Multiple Sclerosis Patients.Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Entsar Karem Abd Elazeem, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCDCS in MS
Record Dates: First submitted 2022-05-18; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Transcranial direct current stimulation; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial-controlled study to assess the ability of tDCS; anodal stimulation of left DLPC versus sham stimulation in improving fatigue in MS patients
Who Masked: Participant, Investigator
Masking Description: Anodal, or sham with a ratio 1:1 were placed in serially numbered opaque closed envelopes. Each patient was given a serial number from a computer generated randomization table, and was placed in the appropriate group after opening the corresponding sealed envelope.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Participants in the experimental groups received ten -sessions a-tDCS (1.5mA, 20minutes) anodal stimulation of left DLPC over two weeks duration (five sessions per week).
  Interventions: Device: a-tDCS
- sham group (Sham Comparator): The sham group received ten sessions of sham stimulation for 20-minutes in each session.
  Interventions: Device: a-tDCS

INTERVENTIONS:
Device: a-tDCS — Transcranial direct current stimulation

SUMMARY:
This work is aimed to assess the long term effect of TDCS in fatigue management among MS patients

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an inflammatory demyelinating disease of the central nervous system that is considered one of the most frequent causes of disability in the young adult.

Fatigue in MS may affect up to 80 % of the people with MS. It tends to persist over time once it appears. However, despite high frequency, fatigue remains poorly understood. Fatigue in MS is neither consistently linked to disease severity nor disease duration, although it is found to be worse in individuals with the secondary progressive subtype.

Fatigue is distinct from sleepiness, and fails to improve with adequate sleep. Multiple factors are thought to contribute to fatigue[7 , 8] with no specific biomarker or etiology yet confirmed.

A wide variety of therapies have been tested to reduce fatigue in MS, but unfortunately, none have been consistently effective. Transcranial direct current stimulation (tDCS) is a relatively recent therapeutic development that utilizes low-amplitude direct currents to induce changes in cortical excitability. Although various non-invasive neuromodulation technologies are available , tDCS has unique advantages compared to other stimulation methods such as its ease of use, lower cost, and greater safety and tolerability.

Small preliminary studies have observed that tDCS may be a promising treatment for MS fatigue, using sham-controlled crossover designs, with five tDCS sessions, using either a motor, sensory, or dorsolateral prefrontal cortex (DLPFC). Recently Chalah et al.[12] study demonstrated that DLPFC (left anodal) when compared the posterior parietal cortex led to the most fatigue specific improvements.

Thus, tDCS can reduce fatigue burden for people with MS, it may be possible to implement a tDCS therapy for symptomatic management of fatigue.

ELIGIBILITY:
Inclusion Criteria:

Any adult patient will be fulfilling diagnostic criteria of Multiple sclerosis and could be providing consent for participation in the study, will be included in the study.

Exclusion Criteria:

* any patient showed this following condition will be excluded from the study;
* Any MS patient had any contraindication condition to use TMS or TCDS (such as epilepsy, head trauma, metallic procedure, cerebral insult)
* Any patient had infection or febrile condition.
* Any patient had other co morbid neurological or psychiatric disorders or systemic disease.
* Any patient refuses participation in study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
fatigue assessment scale | at post sessions, 1 month and 2 month post sessions
  it is a acale filed by the patient and it consists of scale from 1 to 10
visual analogue scale | at post sessions, 1 month and 2 month post sessions
  it is a scale from 0 to 10 to assess major fatigue

SECONDARY OUTCOMES:
changes in cortical excitability parameters at post 10th session compared to baseline measurements of cortical excitability parameters | at post sessions, 1 month and 2 month post sessions
  Detection of the relationship between cortical excitability changes{after 10th session) and changes in fatigue and HDS and QLoL changes..

CONTACTS AND LOCATIONS:
Overall Officials: Noha M Abo-Elfetoh, PHD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- See also: Compston A, Coles A. Multiple sclerosis. Lancet. — http://www.proquest.com/openview/adf0bd26e1b74ed3eeec5d8453bb657e/1?cbl=2029739&pq-origsite=gscholar&parentSessionId=D5TfE0n2xAVp%2F3af%2BtR8AsLlrvRjuA2r5I7x%2Bj%2BymuI%3D
- See also: Tellez N et al. Fatigue in multiple sclerosis persists over time: a longitudinal study. J Neurol — http://link.springer.com/article/10.1007/s00415-006-0247-3
- See also: Krupp L. Fatigue is intrinsic to multiple sclerosis (MS) and is the most commonly reported symptom of the disease. Mult Scler — https://pubmed.ncbi.nlm.nih.gov/16900749/
- See also: Ghajarzadeh M, Jalilian R, Eskandari G, et al. Fatigue in multiple sclerosis: Relationship with disease duration, physical disability, disease pattern, age and sex. Acta Neurol Belg — http://link.springer.com/article/10.1007/s13760-013-0198-2
- See also: Chen MY, Wang EK, Jeng YJ. Adequate sleep among adolescents is positively associated with health status and health-related behaviors. BMC Public Health — http://bmcpublichealth.biomedcentral.com/articles/10.1186/1471-2458-6-59
- See also: Genova HM, Rajagopalan V, Deluca J, et al. Examination of cognitive fatigue in multiple sclerosis using functional magnetic resonance imaging and diffusion tensor imaging. PLoS ONE. — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0078811
- See also: Generalizing remotely supervised transcranial direct current stimulation (tDCS): feasibility and benefit in Parkinson's disease — https://link.springer.com/article/10.1186/s12984-018-0457-9
- See also: Multi-session anodal transcranial direct current stimulation enhances lower extremity functional performance in healthy older adults — https://link.springer.com/article/10.1007/s00221-020-05827-6